CLINICAL TRIAL: NCT01909596
Title: Does it Exist a Relationship Between Inclination Angle of Foot Orthoses and Varus Angle of the Knee in the Relief of the Knee Osteoarthritis Symptoms?
Brief Title: Lateral Wedge Insoles With Arch Support in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Fonds de la Recherche en Santé du Québec (Other Government); Ergorecherche Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OP-2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-26 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Medial Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Knee osteoarthritis patients - No insoles (No Intervention): Without orthoses
- Knee osteoarthritis patients - Customised (Active Comparator): Medial arch support without lateral wedge
  Interventions: Device: Neutral customized foot orthoses
- Knee osteoarthritis patients - Customised + 6° (Active Comparator): 6° lateral wedge insoles + Medial arch support
  Interventions: Device: 6° lateral customized foot orthoses
- Knee osteoarthritis patients - Customised + 10° (Active Comparator): 10° lateral wedge insoles + Medial arch support
  Interventions: Device: 10° lateral customized foot orthoses

INTERVENTIONS:
Device: Neutral customized foot orthoses — Foot orthoses with arch support and without lateral inclination
  Other Names: Orthoconcept Inc, Laval, Qc, Canada
  Arms: Knee osteoarthritis patients - Customised
Device: 6° lateral customized foot orthoses — Foot orthoses with arch support above insoles with lateral inclination set at 6°
  Other Names: Orthoconcept Inc, Laval, Qc, Canada
  Arms: Knee osteoarthritis patients - Customised + 6°
Device: 10° lateral customized foot orthoses — Foot orthoses with arch support above insoles with lateral inclination set at 10°
  Other Names: Orthoconcept Inc, Laval, Qc, Canada
  Arms: Knee osteoarthritis patients - Customised + 10°

SUMMARY:
The purpose of this is to test lateral foot orthoses with different amount of wedging to find a model that predicts the optimal lateral inclination of foot orthosis based on biomechanical or feelings measures. This study was a cross-sectional study with patients serving as their own control. The investigators recruited 24 knee osteoarthritis. Knee radiography and clinical angles measures was carried out before making orthoses, then motion analysis with an optoelectronic system was performed with each pair of foot orthoses. During motion analysis, five gait trials were carried out in each condition.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial knee osteoarthritis (OA ; Kellgren-Lawrence grade I, II or III) according to clinical and radiological criteria of the American College of Rheumatology
* Knee pain > 31/100 (Western Ontario and McMaster Universities Arthritis Index - WOMAC)
* Moderately active
* Varus knee alignment equal or superior to 2°

Exclusion Criteria:

* Severe knee OA (K-L grade IV)
* Rheumatoid arthritis or other inflammatory arthritis
* Avascular necrosis
* History of periarticular fracture or septic arthritis
* Bone metabolic disease
* Pigmented villonodular synovitis
* Cartilaginous disease
* Neuropathic arthropathy
* Synovial osteochondromatosis
* Total or partial knee arthroplasty
* Flexion contracture of ipsi- or contra-lateral knee greater than 15°
* Hip or ankle joint damage with mobility limitation
* Obesity (BMI ≥ 40)
* Intra-articular corticosteroids injection in the affected knee during the two previous months
* Reduced mobility (Charnley class C)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Knee pain | At time of device receipt
  A 20-cm visual analog scale (0-100) is used to assess pain.
Knee adduction moment | At time of device receipt
  Measure of the knee adduction moment is a non invasive technic to identify change in medial knee loading, major problem in medial knee osteoarthritis.

SECONDARY OUTCOMES:
Foot orthoses comfort | At time of device receipt
  A 20-cm visual analog scale (0-100) is used to assess comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, PhD, Study Director — Laval University; Yoann Dessery, MSc, Principal Investigator — Laval University; Étienne L Belzile, MD, Study Director — Laval University
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Quebec, Canada